CLINICAL TRIAL: NCT02086474
Title: Daily Activity Quantification and Gait Pattern Analysis Before and After Intra-articular Injection of Viscosupplement Among Hip Osteoarthritis Patients
Brief Title: Daily Activity and Gait Analysis After Viscosupplement Injection Among Hip Osteoarthritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Philippe Corbeil, PhD, Laval University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INF-2014
Record Dates: First submitted 2014-03-07; First posted 2014-03-13 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Hyaluronic Acid; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyaluronan (Experimental): Hyaluronan acid Neovisc : one 6cc (viscosupplement) intra-articular injection
  Interventions: Drug: Hyaluronan
- Bupivacaine (Placebo Comparator): one Marcain extra-capsular injection
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Hyaluronan — Intra-articular injection
  Other Names: Hyaluronan acid : Neovisc®
  Arms: Hyaluronan
Drug: Bupivacaine — Extra-capsular injection
  Other Names: Bupivacaine: Marcaine®
  Arms: Bupivacaine

SUMMARY:
The objective of this study is to assess the changes in daily physical activity and gait pattern, following a viscosupplement injection among a population who is suffering from hip osteoarthritis. A kinetic and kinematic gait analysis, an Actigraph activity monitor, a functional Timed-Stair-Test and two questionnaires (Medical Outcome Study Short-Form36 (MOS-SF36), Hip disability and Osteoarthritis Outcome Score (HOOS)) about how the pathology affects the quality of life, will be use.

ELIGIBILITY:
Inclusion Criteria:

* From 45 years old to 65 years old
* Clinically symptomatic moderate or severe hip osteoarthritis (Tönnis Grade II to III)
* Capacity to keep steady upright position and walking during 15 minutes
* Body mass index < 40kg/m2

Exclusion Criteria:

* Bilateral hip osteoarthritis
* No broken hip or leg during the last 12 months
* Bone necrosis
* Rheumatoid arthritis, articular chondrocalcinosis, metabolic bone disease, psoriasis, gout, active infection
* Per os corticosteroid treatment
* Corticosteroid injection < 3 months
* Viscosupplement injection < 6 months
* Hypersensitivity to hyaluronic acid products
* Planed surgery during study duration
* Physical or mental disability to fill in questionnaires and/or to participate to follow-up

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change in hip flexion-extension range of motion | Change from Baseline at 6 months
  Subtraction between maximum and minimum flexion measured with motion capture system during gait
Change in daily physical activity | Change from Baseline at 6 months
  Intensity and duration of the daily physical activity measured with pedometer

SECONDARY OUTCOMES:
Change in hip pain | change from Baseline at 6 months
  Questionnaires HOOS
Change in quality of life | Change from Baseline at 6 months
  Questionnaires: MOS-SF36 and HOOS
Change in walking cadence | Change from Baseline at 6 months
  Measured during 3D gait analysis

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Cantin-Warren, B.Sc., Principal Investigator — Laval University; Étienne L. Belzile, MD, Study Director — Laval University; Philippe Corbeil, Ph.D., Study Director — Laval University
Locations (1):
- Pavillon de l'Éducation Physique et des Sports - Université Laval, Québec, Canada